CLINICAL TRIAL: NCT00729703
Title: Optimal Antitachycardia Therapy in ICD Patients Without Pacing Indications
Brief Title: Optimal Anti-tachycardia Therapy in Implantable Cardioverter-defibrillator (ICD) Patients Without Pacing Indications
Acronym: OPTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPTION - ITAC03
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Tachycardia
Keywords: ICD; Minimized; ventricular; pacing; indication; Clinical outcome; Inappropriate shock
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dual-chamber detection and activated treatment (at least ATP) in the slow VT-zone plus activated AAIsafeR pacing (basic rate 60 bpm).
  Interventions: Device: Ovatio DR 6550
- 2 (Experimental): Single-chamber ICD following clinical practice but with a monitoring zone active to allow the documentation of all occurring ventricular arrhythmias
  Interventions: Device: OVATIO DR 6550

INTERVENTIONS:
Device: Ovatio DR 6550 — Dual-chamber ICD therapy with minimized ventricular pacing
  Arms: 1
Device: OVATIO DR 6550 — Single-chamber device therapy with settings which are common in clinical practice.
  Arms: 2

SUMMARY:
This study evaluates the impact of a new pacing mode avoiding unnecessary ventricular stimulation in combination with advanced dual chamber detection with slow VT management on the clinical outcome for hospitalization and mortality and inadequate therapy in medically stable, ICD-indicated patients with impaired left ventricular function (LVEF ≤ 40%) who do not have pacing indications and no indication for Cardiac Resynchronization Therapy (CRT). It compares a new pacing mode avoiding ventricular stimulation when not needed combined with dual chamber detection with a pure ventricular back up pacing and single chamber detection criteria with pure ventricular back up pacing. Therapies are compared in a prospective, randomized, single-blinded, parallel trial with a 24-month randomized treatment period. Randomization follows a 1:1 ratio. ICD therapy is enabled for all patients throughout the study. All patients receive optimal drug therapy for arrhythmia and heart failure treatment.

DETAILED DESCRIPTION:
All patients will receive an implantable cardioverter defibrillator OVATIO™ DR model 6550 or a later Sorin Group device offering the same functions. After Enrolment visit but before implant, patients will be randomized in two arms according to the parallel study design. Whenever possible before implant there will be the first Holter recording for the Tvar risk stratification procedure. In case Tvar recording could not be performed before implant it has to be performed before patient leaves the hospital post implant in unpaced rhythm.

The dual-chamber arm will be programmed to 3 detection zones with PARAD+ activated.

The TDI for the slow VT zone will be set to 500 ms (120 bpm - or in case the resting rate is higher than 90 bpm it is recommended to adjust this parameter to: resting rate + 30 bpm) and at least one ATP program activated as specified in table 1.

A VT zone with a TDI of 353 ms (170 bpm) in case of no history of VT or a TDI cycle length equalling slowest documented VT interval (spontaneous or induced) plus 50 ms is required. In this 2nd VT zone therapies need to be activated in this group.

AAIsafeR2 mode will be activated with a basic rate of 60 bpm. The single-chamber arm will be programmed to optimal detection with Acceleration (Onset), Stability and Long Cycle Search (VTLC) activated. A VT zone is requested in this group, with the same programming procedures as described above. Therapies will be set according to the clinical judgment of the participating investigators but a Slow VT-zone with TDI 500 ms in monitoring setting at least is required.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been prescribed the implantation for an ICD system accordingly to the relevant currently-approved ACC/AHA guidelines 1 or ESC guidelines 35 or any relevant currently-approved local guidelines for the implantation of an ICD-system
* Impaired left ventricular function demonstrated by a left-ventricular ejection fraction (LVEF) ≤ 40 %, measured by angio-scintigraphy, echocardiography, or contrast ventriculogram.
* An optimal (as determined by the enrolling physician) medical regimen.
* Patient has received all relevant information on the study, and has signed and dated a consent form.

Exclusion Criteria:

* Any generally accepted indication for standard cardiac pacing, or any contraindication for standard cardiac pacing.
* Any indication for CRT accordingly to the relevant currently-approved ACC/AHA1 or ESC35 guidelines for the implantation of a CRT system.
* Any contraindication for ICD therapy and the implant of a dual chamber ICD.
* ICD replacement
* Chronic atrial arrhythmias or cardioversion for atrial fibrillation within the past month.
* A PR interval > 250 ms or AR interval > 300 ms measured at implant.
* Hypertrophic obstructive cardiomyopathy.
* Acute myocarditis.
* Unstable coronary symptoms or myocardial infarction within the last month.
* Recent (within the last month) or planned cardiac revascularization or coronary angioplasty.
* Recently performed (in the last month) or planned cardiac surgery
* Already included in another clinical study.
* Life expectancy less than 24 months.
* Inability to understand the purpose of the study or refusal to cooperate.
* Inability or refusal to provide informed consent and, if not part of the informed consent, a Health Insurance Portability and Accountability Act (HIPAA) authorization.
* Unavailability for scheduled follow-up at the implanting or cooperating center.
* Age of less than 18 years.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The first part is the time to first occurrence of inappropriate ICD shock therapy. The second part is the composite endpoint of time to first occurrence of death (all causes)or Hospitalizations due to cardio-vascular event. | implant, 3 months, 9 months, 15 months, 21 months and 27 months

SECONDARY OUTCOMES:
all cause mortality and cardio-vascular related mortality | 27 months follow up
Hospitalizations due to cardio-vascular event (specified for each type of event) | 27 months follow up
Time to first occurrence of inappropriate ICD shock therapy | 27 months follow up
Evaluation of the impact of the different therapies on quality of life and heart failure status | 27 months follow up
Sensitivity and specificity for VT/SVT discrimination for the first 100 patients in each group. | 27 months
Inappropriate overall device reactions defined by inappropriate shock and/or ATP therapy or inappropriate therapy delay/inhibition > 2 minutes on VTs | 27 months
time to first documented AF occurrence and number of patients moving into permanent or persistent AF | 27 months follow up
Cardiac dimensions obtained by echo evaluation for a subset of patients of both groups | Baseline and 27 months
Slow VT incidence | 27 months
Unscheduled visits and hospitalizations due to slow VT | 27 months follow up
System related complications including lead dislodgements, exit block, oversensing which requires programming corrections, infections, complications which require reintervention | 27 months follow up
Cumulative percentage of ventricular pacing and proportion of patients with 0% V pacing. | 27 months follow up
Overall success rate of ATP in the FVT zone | 27 months
Cost effectiveness of applied ICD therapy | 27 months
PPV and NPV for Tvar risk stratification | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Kolb, Principal Investigator — Deutsches Herzzentrum München
Locations (55):
- United States (5):
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Atlanta Va Medical Center, Decatur, Georgia
  - Southern Medical Research, Llc, Mandeville, Louisiana
  - River City Cardiology, Jeffersonville, Ohio
  - Pee Dee Cardiology, Florence, South Carolina
- Belgium (3):
  - Algemeen Ziekenhuis - Antwepen, Antwepen
  - Kliniek Maria Middelares - Gent, Ghent
  - Heart Center Virga Jesse Ziekenhuis - Hasselt, Hasselt
- Canada (2):
  - CHUM Hotel-Dieu, Montreal
  - Hôpital Sacré Coeur, Montreal
- France (16):
  - Centre Hospitalier General, Aix-en-Provence
  - CHU Le Haut L'Evêque, Bordeaux
  - CHU Hôpital Michallon Grenoble, Grenoble
  - Clinique De Parly II, Le Chesnay
  - Clinique les sources, Le Mans
  - CH ST Philibert, Lomme
  - Hôpital St Joseph, Lyon
  - Hopital Arnaud De Villeneuve, Montpellier
  - CHU Nantes, Nantes
  - Clinique Bizet, Paris
  - CH Pau, Pau
  - CHU Charles Nicolle, Rouen
  - Clinique Pasteur, Toulouse
  - Hôpital Rangueil, Toulouse
  - CHU Purpan Toulouse, Toulouse
  - CHU Tours, Tours
- Germany (18):
  - Herzkreislaufklinik, Bad Bevensen
  - Kerckhoff Klinik, Bad Nauheim
  - Charite Campus Virchow, Berlin
  - Universitätskliniken Bonn, Bonn
  - Klinikum Coburg, Coburg
  - Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universität des Saarlandes, Homburg
  - Universitatsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Kardiologische Gemeinschaftspraxis, München
  - Universitatsklinikum Grosshadern, München
  - DHZ Munchen, München
  - Klinikum Bogenhausen, München
  - Klinikum rechts der Isar, München
  - Uniklinik Munster, Münster
  - Klinikum der Universität Regensburg, Regensburg
  - Krankenhaus der Barmherzigen Brüder, Regensburg
  - Universitätsklinik Ulm, Ulm
- Italy (5):
  - Ospedale Civile, Desio
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Casa Di Cura Citta Di Pavia, Pavia
  - Policlinico San Donato, San Donato
  - Ospedale Clinicizzato San Donato, San Donato Milanese
- Onze Lieve Vrouwen Gasthuis, Amsterdam, Netherlands
- Portugal (2):
  - Hospital Garcia de Orta, Almada
  - Hospital Senhora da Oliveira, Guimarães
- United Kingdom (3):
  - St Peters Hospital, London
  - Musgrove Park Hospltal, Taunton
  - Worthing And Southlands Hospital, Worthing

REFERENCES:
- [Background] Kolb C, Tzeis S, Sturmer M, Babuty D, Schwab JO, Mantovani G, Janko S, Aime E, Ocklenburg R, Sick P. Rationale and design of the OPTION study: optimal antitachycardia therapy in ICD patients without pacing indications. Pacing Clin Electrophysiol. 2010 Sep;33(9):1141-8. doi: 10.1111/j.1540-8159.2010.02790.x. PMID 20487351
- [Result] Kolb C, Sturmer M, Sick P, Reif S, Davy JM, Molon G, Schwab JO, Mantovani G, Dan D, Lennerz C, Borri-Brunetto A, Babuty D. Reduced risk for inappropriate implantable cardioverter-defibrillator shocks with dual-chamber therapy compared with single-chamber therapy: results of the randomized OPTION study. JACC Heart Fail. 2014 Dec;2(6):611-9. doi: 10.1016/j.jchf.2014.05.015. Epub 2014 Oct 1. PMID 25282033